CLINICAL TRIAL: NCT01255215
Title: Inhaled Nitric Oxide for the Adjunctive Therapy of Severe Malaria: a Randomized Controlled Trial
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Collaborators: Makerere University (Other); University of Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: iNO RCT
Record Dates: First submitted 2010-12-05; First posted 2010-12-07 (Estimated); Last update posted 2014-02-20 (Estimated); Status verified 2012-12

CONDITIONS: Severe Malaria
Keywords: malaria; children
MeSH Terms: conditions — Malaria | interventions — Nitric Oxide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Inhaled Nitric Oxide (Experimental): iNO, a gaseous molecule, will be administered by inhalational route over a maximum period of 72 hours.
  Interventions: Drug: Inhaled Nitric Oxide
- Room air (Placebo Comparator): Room air will be delivered by air compressor through an indistinguishable mask system.
  Interventions: Drug: Inhaled Nitric Oxide

INTERVENTIONS:
Drug: Inhaled Nitric Oxide — Form: Gas (inhalational) Dose: 80 ppm Dosing schedule: Continuous Treatment period: Maximum 72 hours (may be discontinued earlier if patient recovers and no longer tolerates face mask)
  Other Names: NO, nitrogen monoxide

SUMMARY:
Despite the use of highly effective anti-malarial medications, 10-30% of African children with severe malaria will die, underscoring the need for adjunctive therapies that can be applied in endemic areas. A clinical trial of adjunctive inhaled nitric oxide (iNO) in severe malaria is warranted on the basis of firm proof of concept from animal studies and a human study using the NO donor L-arginine, together with evidence of safety from clinical experience and trials of iNO for other conditions. Our objective is to determine whether supplemental iNO (80 ppm) in addition to Ugandan Standard of Care treatment reduces levels of Angiopoietin-2 (Ang-2), a quantitative biomarker of malaria severity, in children with severe malaria compared to Standard of Care treatment alone. We will conduct a randomized placebo-controlled trial among children 1-10 years of age admitted to Jinja Hospital (Uganda) with severe malaria to test the efficacy of inhaled nitric oxide in severe malaria.

DETAILED DESCRIPTION:
Severe malaria remains a major cause of global morbidity and mortality. While the use of artemisinin-based antimalarial therapy has improved outcomes in severe malaria, the mortality rate remains high. Adjunctive therapies that target the underlying pathophysiology of severe malaria may further reduce morbidity and mortality. Endothelial activation plays a central role in the pathogenesis of severe malaria, of which the angiogenic factors angiopoietin-1 (Ang-1) and angiopoietin-2 (Ang-2) have recently been shown to function as key regulators. Nitric oxide (NO) is a major inhibitor of Ang-2 release from endothelium and has been shown to decrease endothelial inflammation and reduce the adhesion of parasitized erythrocytes. Low-flow inhaled nitric oxide gas (iNO) is a US FDA-approved treatment for hypoxic respiratory failure in neonates. Based on compelling data on the efficacy of iNO in experimental cerebral malaria in animal models, coupled with the documented safety of iNO in clinical practice and trials for other diseases, we propose a randomized clinical trial of iNO for the adjunctive treatment of severe malaria in Ugandan children.

ELIGIBILITY:
Inclusion Criteria:

* Age 1-10 years
* Positive malaria rapid diagnostic test in the presence of any of the features of severe malaria
* Willing and able to complete follow up schedules for the study - 14 day and 6 months after hospital discharge

Exclusion Criteria:

* Baseline methemoglobinemia
* Known renal, cardiac, or hepatic disease or other chronic illnesses like diabetes, epilepsy, cerebral palsy, clinical AIDS
* Severe malnutrition
* Severe malarial anemia without other signs of severe malaria

Ages: 1 Year to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 180 (Actual)
Dates: Start 2011-07; Primary Completion 2013-07 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Change in serum angiopoietin-2 level | Admission through 72 hours
  Daily Ang-2 measurements over the first 72 hours of hospital admission will be the primary efficacy outcome. Elevated Ang-2 levels are associated with poor clinical outcome in severe malaria and Ang-2 has been used to follow disease progression and recovery in previous studies of malaria. Thus, Ang-2 is an objective, quantitative surrogate marker of disease severity, validated for longitudinal follow-up of patients with malaria.

SECONDARY OUTCOMES:
Mortality | 48 hours and 14 days after admission
Time to hospital discharge | From admission to approximately 72 hours
  Recovery times (time to fever resolution, time to sit unsupported, and time to hospital discharge) are standard, clinically relevant outcomes in other therapeutic trials for malaria.
Time to parasite clearance. | From admission to approximately 72 hours
  Parasitological efficacy outcome; quantitative assessment of parasite density by light microscopy of Giemsa-stained thin smears.
Biomarkers and genetic determinants of endothelial activation, inflammation and coagulopathy, to be determined. | From admission to approximately 72 hours
  Biomarkers and genetic determinants of severe malaria pathogenesis may provide additional insight into the pathways and processes altered in cerebral malaria and affected by iNO delivery. We plan to examine biomarkers of endothelial activation, inflammation including cytokines, and coagulopathy which are central to the pathophysiology of severe malaria. In addition, genetic pathways involved in severe malaria and response to iNO will be investigated.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Hawkes, MD, Study Director — University of Toronto
Locations (1):
- Jinja Regional Referral Hospital, Jinja, Uganda

REFERENCES:
- [Result] Neonatal Inhaled Nitric Oxide Study Group. Inhaled nitric oxide in full-term and nearly full-term infants with hypoxic respiratory failure. N Engl J Med. 1997 Feb 27;336(9):597-604. doi: 10.1056/NEJM199702273360901. PMID 9036320
- [Result] Davidson D, Barefield ES, Kattwinkel J, Dudell G, Damask M, Straube R, Rhines J, Chang CT. Inhaled nitric oxide for the early treatment of persistent pulmonary hypertension of the term newborn: a randomized, double-masked, placebo-controlled, dose-response, multicenter study. The I-NO/PPHN Study Group. Pediatrics. 1998 Mar;101(3 Pt 1):325-34. doi: 10.1542/peds.101.3.325. PMID 9480993
- [Result] Dobyns EL, Cornfield DN, Anas NG, Fortenberry JD, Tasker RC, Lynch A, Liu P, Eells PL, Griebel J, Baier M, Kinsella JP, Abman SH. Multicenter randomized controlled trial of the effects of inhaled nitric oxide therapy on gas exchange in children with acute hypoxemic respiratory failure. J Pediatr. 1999 Apr;134(4):406-12. doi: 10.1016/s0022-3476(99)70196-4. PMID 10190913
- [Result] Michael JR, Barton RG, Saffle JR, Mone M, Markewitz BA, Hillier K, Elstad MR, Campbell EJ, Troyer BE, Whatley RE, Liou TG, Samuelson WM, Carveth HJ, Hinson DM, Morris SE, Davis BL, Day RW. Inhaled nitric oxide versus conventional therapy: effect on oxygenation in ARDS. Am J Respir Crit Care Med. 1998 May;157(5 Pt 1):1372-80. doi: 10.1164/ajrccm.157.5.96-10089. PMID 9603111
- [Result] Dellinger RP, Zimmerman JL, Taylor RW, Straube RC, Hauser DL, Criner GJ, Davis K Jr, Hyers TM, Papadakos P. Effects of inhaled nitric oxide in patients with acute respiratory distress syndrome: results of a randomized phase II trial. Inhaled Nitric Oxide in ARDS Study Group. Crit Care Med. 1998 Jan;26(1):15-23. doi: 10.1097/00003246-199801000-00011. PMID 9428538
- [Result] Troncy E, Collet JP, Shapiro S, Guimond JG, Blair L, Ducruet T, Francoeur M, Charbonneau M, Blaise G. Inhaled nitric oxide in acute respiratory distress syndrome: a pilot randomized controlled study. Am J Respir Crit Care Med. 1998 May;157(5 Pt 1):1483-8. doi: 10.1164/ajrccm.157.5.9707090. PMID 9603127
- [Result] Lundin S, Mang H, Smithies M, Stenqvist O, Frostell C. Inhalation of nitric oxide in acute lung injury: results of a European multicentre study. The European Study Group of Inhaled Nitric Oxide. Intensive Care Med. 1999 Sep;25(9):911-9. doi: 10.1007/s001340050982. PMID 10501745
- [Result] Gerlach H, Keh D, Semmerow A, Busch T, Lewandowski K, Pappert DM, Rossaint R, Falke KJ. Dose-response characteristics during long-term inhalation of nitric oxide in patients with severe acute respiratory distress syndrome: a prospective, randomized, controlled study. Am J Respir Crit Care Med. 2003 Apr 1;167(7):1008-15. doi: 10.1164/rccm.2108121. PMID 12663340
- [Result] Taylor RW, Zimmerman JL, Dellinger RP, Straube RC, Criner GJ, Davis K Jr, Kelly KM, Smith TC, Small RJ; Inhaled Nitric Oxide in ARDS Study Group. Low-dose inhaled nitric oxide in patients with acute lung injury: a randomized controlled trial. JAMA. 2004 Apr 7;291(13):1603-9. doi: 10.1001/jama.291.13.1603. PMID 15069048
- [Derived] Conroy AL, Hawkes MT, Elphinstone R, Opoka RO, Namasopo S, Miller C, John CC, Kain KC. Chitinase-3-like 1 is a biomarker of acute kidney injury and mortality in paediatric severe malaria. Malar J. 2018 Feb 15;17(1):82. doi: 10.1186/s12936-018-2225-5. PMID 29448936
- [Derived] Bangirana P, Conroy AL, Opoka RO, Hawkes MT, Hermann L, Miller C, Namasopo S, Liles WC, John CC, Kain KC. Inhaled nitric oxide and cognition in pediatric severe malaria: A randomized double-blind placebo controlled trial. PLoS One. 2018 Jan 25;13(1):e0191550. doi: 10.1371/journal.pone.0191550. eCollection 2018. PMID 29370261
- [Derived] Conroy AL, Hawkes M, Hayford K, Hermann L, McDonald CR, Sharma S, Namasopo S, Opoka RO, John CC, Liles WC, Miller C, Kain KC. Methemoglobin and nitric oxide therapy in Ugandan children hospitalized for febrile illness: results from a prospective cohort study and randomized double-blind placebo-controlled trial. BMC Pediatr. 2016 Nov 4;16(1):177. doi: 10.1186/s12887-016-0719-2. PMID 27814710
- [Derived] Hawkes MT, Conroy AL, Opoka RO, Hermann L, Thorpe KE, McDonald C, Kim H, Higgins S, Namasopo S, John C, Miller C, Liles WC, Kain KC. Inhaled nitric oxide as adjunctive therapy for severe malaria: a randomized controlled trial. Malar J. 2015 Oct 29;14:421. doi: 10.1186/s12936-015-0946-2. PMID 26510464
- [Derived] Hawkes M, Opoka RO, Namasopo S, Miller C, Thorpe KE, Lavery JV, Conroy AL, Liles WC, John CC, Kain KC. Inhaled nitric oxide for the adjunctive therapy of severe malaria: protocol for a randomized controlled trial. Trials. 2011 Jul 13;12:176. doi: 10.1186/1745-6215-12-176. PMID 21752262
- [Derived] Hawkes M, Opoka RO, Namasopo S, Miller C, Conroy AL, Serghides L, Kim H, Thampi N, Liles WC, John CC, Kain KC. Nitric oxide for the adjunctive treatment of severe malaria: hypothesis and rationale. Med Hypotheses. 2011 Sep;77(3):437-44. doi: 10.1016/j.mehy.2011.06.003. Epub 2011 Jul 13. PMID 21745716